CLINICAL TRIAL: NCT01915745
Title: Evaluation of the Efficacy of a Mobile Phone Short Message Service on Post-fracture Management for Patients Who Consult to the Emergency Department
Brief Title: Study of Current Practice Evaluating the Efficacy of a Mobile Short Message Service (SMS) on Post-fracture Management.
Acronym: Ostéo-SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K120601; 2012-A01135-38 (Other: European Union Drug Regulatory Authorities Clinical Trial System)
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Low Trauma Non Vertebral Fracture
Keywords: Osteoporosis; Bone densitometry; Fracture; Anti-osteoporotic treatment; Short message service
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usually health care (No Intervention): 85 patients receive the usually health care. Then they are called during 10 minutes at 6 months to check if bone densitometry will be performed and if antiosteoporotic treatment will be initiated.
- Short Message Service - SMS (Experimental): 85 patients receive 3 SMS (at 15 days, 5 weeks and 3 months) after consulting in the Emergency Department emergencies. Then they are called during 10 minutes at 6 months to check if bone densitometry will be performed and if antiosteoporotic treatment will be initiated.
  Interventions: Other: Use of SMS

INTERVENTIONS:
Other: Use of SMS — Patients receive 3 SMS (at 15 days, 5 weeks and 3 months) after consulting in Emergency Department. Then they are called during 10 minutes at 6 months to check if bone densitometry will be performed and if antiosteoporotic treatment will be initiated.
  Other Names: Sending of 3 SMS to remind to the patient to perform bone densitometry.
  Arms: Short Message Service - SMS

SUMMARY:
The purpose of the study is to show that the standardized sending of SMS improve the bone mineral density (BMD) screening of patients seen in the Emergency department for low trauma fracture.

DETAILED DESCRIPTION:
Osteoporosis is a significant health problem in the older population affecting at least 40% of women and 15 % of men over the age of 50 years. Fracture leads to increased morbidity and mortality and healthcare costs as well as predisposing to future fractures. Patients with a history of low-energy fracture are at significantly increased risk for further fractures in the short-term. There is a universal consensus supported by high-quality randomized trial evidence for secondary prevention: patients with low-trauma fragility fractures should have BMD testing and most of them would benefit from anti-osteoporotic treatment There is, unfortunately, also a well-documented and near-universal gap between evidence-based best practice and usual care for patients with fragility fractures. Although osteoporotic fracture indicates a two- to threefold increased risk of future fracture, only one in five patients receive medical intervention after sustaining an osteoporotic fracture. Diverse post fracture interventions have been developed for improving osteoporosis diagnosis and treatment: provided educational materials to patients and/or primary physician, use of medical reminders, more intensive interventions using osteoporosis case manager (nurse, doctor) and fracture liaison service. the most effective post fracture interventions are those which are more proactive, complex, time consuming, coordinator manager dependant, and costly. Taking account the costs and the humans resources needing, we propose to improve post fracture patient management using mobile telecommunication already used for other chronic diseases management. There is no study about the use of phone short message service (SMS) support in the field of osteoporosis, especially in the post-fracture management: bone mineral density (BMD) screening, anti-osteoporotic treatment initiation and monitoring and improvement of adherence. One of the limitations could be the use of phone mobile in these older patients. We assessed the number of mobile phone users among 100 consecutive subjects who were hospitalized for non vertebral fracture (mean age 69.5 years (50-98); 58 women and 42 men) in the Emergency department of Cochin hospital: 61 % had a mobile phone and used SMS; 61% have a mobile phone.

We propose to assess the efficacy of the use of SMS support to improve the screening and the initiation of antiosteoporotic treatment in patients with low trauma non vertebral fracture, who consult in Emergency department.

This is a study of current care, monocentric, randomized, open. 170 patients will be followed for 6 months. The group control will receive the usual recommendations to make an appointment of realization of bone densitometry. The SMS group will receive 3 SMS (at 15 days, 5 weeks and 3 months) after consulting the time of consultation in Emergency department, and will be called during 10 minutes at 6 months by a nurse.

The results of this study will have an important impact for the postfracture management in the field of osteoporosis . Indeed, if we demonstrate that the use of SMS improves the BMD screening and antiosteoporotic treatment initiation, we plan to assess in a large randomized controlled trial whether mobile phone communication can decrease the risk of new fracture comparatively to usual care in patients with low trauma fracture could use.

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 50 years old
* Low trauma non vertebral fracture
* Ambulatory patient
* Direct access to mobile phone (or access with the help of a close person) and ability to communicate via SMS.
* Patient who doesn't oppose to his participation in the study
* Affiliation to the social security

Exclusion Criteria:

* Patients hospitalized for the fracture in the orthopaedics department because these more severe patients have a systematic screening and management of osteoporosis.
* Fractures whose location is not suggestive of osteoporotic fracture (cervical spine, skull, hands, fingers, toes)
* Pathological fractures (cancer or myeloma)
* Traumatic fractures
* Severe alterations of cognitive functions
* Resident subjects except Paris and the surrounding area

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Realisation of bone densitometry | 6 months
  Realisation of a bone densitometry within 6 months after the consultation in the Emergency Department

SECONDARY OUTCOMES:
The initiation of a treatment anti-osteoporotic | 6 months
  Initiation of a treatment anti-osteoporotic (calcium and/or vitamine D, raloxifene, bisphosphonates, teriparatide, ranelate de strontium, denosumab) within 6 months after the consultation in the Emergency Department for low trauma fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Karine BRIOT, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Hospital Cochin, Paris, France